CLINICAL TRIAL: NCT06826625
Title: Elucidation of the Oxidative Mechanism Effective in Polycystic Ovary Syndrome: a Randomized Controlled Clinical Study
Brief Title: Oxidative Stress in Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, Hasan Basri Savas, Associate Professor, Mardin Artuklu University
Other Study IDs: 2020/23-11
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Polycystic Ovarian Syndrome (PCOS); Oxidative Stress
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- polycystic ovary syndrome: Woman with PCOS
- control: Women without PCOS

SUMMARY:
The aim of the study was to determine changes in hematological and biochemical parameters and specific oxidative stress markers in patients with PCOS.

ELIGIBILITY:
Inclusion Criteria:

The PCOS group included patients with oligomenorrhea (menstrual period intervals of more than 35 days), clinical signs of hyperandrogenism (acne or hirsutism), biochemical signs of hyperandrogenism (with total testosterone of 100 ng/dL and above and patients with dehydroepiandrosterone sulfate of 400 g/dl and above), an LH/FSH ratio of over 3 on the second day of the menstrual period, a body mass index of 25 and above, and polycystic ovaries detected in suprapubic ultrasonography.

Exclusion Criteria:

Pregnant individuals, individuals with diabetes mellitus, metabolic syndrome, adrenal pathology, pelvic mass, and malignancy were not included in the study.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Woman with and without polycystic ovary syndrome
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Oxidative stress markers | From January 2021 to December 2021
  TAS, TOS, OSI, PON, ARES, total thiol, native thiol, disulfide (-S-S-), reduced thiol, oxidized thiol, and IMA

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Training and Research Hospital Gynecology and Obstetrics Department, Antalya, Turkey (Türkiye)